CLINICAL TRIAL: NCT05604495
Title: The Clinical and Genetic Characteristics of Cystic Fibrosis and Cystic Fibrosis Disorders in Chinese Adults With Bronchiectasis
Brief Title: Screening for Cystic Fibrosis and Cystic Fibrosis Related Disorders in Chinese Adults With Bronchiectasis
Status: Recruiting | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Jin-Fu Xu, Director, Head of respiratory medicine, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: 20220922
Record Dates: First submitted 2022-10-25; First posted 2022-11-03 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Cystic Fibrosis, Pulmonary
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Genomic DNA extracted from peripheral whole blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with bronchiectasis (unknown cause): Diagnosis of bronchiectasis was performed using chest HRCT scans in suspected patients with coughing and expectoration, or long durations of hemoptysis. High-resolution images were obtained during full inspiration at 1-mm collimation and 10-mm intervals from the apex to the base of the lungs. The presence of bronchiectasis was confirmed based on the following criteria: 1) lack of tapering in the bronchi; 2) dilation of the bronchi where the internal diameter was larger than that of the adjacent pulmonary artery; or 3) visualization of the peripheral bronchi within 1 cm of the costal pleural surface or the adjacent mediastinal pleural surface.
  Interventions: Diagnostic Test: Sweat Test

INTERVENTIONS:
Diagnostic Test: Sweat Test — In people with cystic fibrosis (CF), there is a problem in the transport of chloride across cell membranes. This results in higher concentrations of chloride (as salt) in sweat compared to those who do not have cystic fibrosis. So, if there is a family history or a possibility of CF, the sweat test is part of the special tests to help make, or exclude, a diagnosis of cystic fibrosis.

SUMMARY:
The study carries out Sweet Tests and CFTR-mutation screening to explore the prevalence, clinical characteristics, and prognosis of cystic fibrosis, as well as the CFTR-mutation spectrum in Chinese adults with bronchiectasis. The study is multi-centered, prospective, non-interventional, and observational.

DETAILED DESCRIPTION:
The incidence of cystic fibrosis (CF) or CFTR dysfunction in China remains unclear due to the absence of a diagnosis and different genetic backgrounds. However, the CF case rate in western countries is relatively high, up to 1/2500. According to the limited statistics, the most common classic clinical symptom of Chinese CF patients is bronchiectasis. Other symptoms often seen in diseased western groups, such as pancreatic insufficiency, are rarely seen in Chinese patients. Thus, Chinese CF or CFTR dysfunction patients easily misdiagnose bronchiectasis, Chronic pneumonia, asthma, etc. Sweet test and CFTR-mutation screening are urgently needed for diagnosing and treating CF or CFTR dysfunction patients in Chinese adults with bronchiectasis. The study will focus on the change in CFTR function, genetic susceptibility factors, and disease progression to explore the incidence, clinical characteristics, and prognosis of cystic fibrosis, as well as the CFTR mutation spectrum in Chinese adults with bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years, the diagnosis of bronchiectasis needs a reference to the definition of "non-cystic fibrosis bronchiectasis guideline" published by the British Thoracic Society in 2017 or 2021 China bronchiectasis expert consensus, clinical symptoms of cough and expectoration, with or without intermittent hemoptysis, and chest CT showed bronchiectasis
* Patients who are willing to sign the consent form and participate in the study.

Exclusion Criteria:

* Patients with incomplete essential information, which is needed for the integrity of data analysis. Essential information includes CT images, respiratory sample cultures, spirometry, and exacerbation history for at least one year.
* Patients under 18 years old.

Sweat Test Exclusion Criteria:

* Patients with an implanted device, such as a defibrillator, neurostimulator, pacemaker, or ECG monitor.
* Patients with a history of epilepsy or seizures.
* Patients who are pregnant.
* Patients that have a known sensitivity or allergy to any ingredient.
* Over-damaged, denuded skin or other recent scar tissue.
* Patients with Cardiac Conditions or with suspected heart problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient recruitment relies on the China Bronchiectasis Registry and Research Collaboration. The final study population will be dynamically adjusted according to the incidence of CF in Chinese adults with bronchiectasis, which will be concluded by the primary study conducted on 200 bronchiectasis patients. 1000 bronchiectasis patients are temporarily decided to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Sweat chloride and conductivity | within 14 days after sweat collection
  Sweat chloride and conductivity is the measured analyte most directly related to the abnormal function of the cystic fibrosis transmembrane regulator (CFTR), the chloride channel that is defective in cystic fibrosis patients

SECONDARY OUTCOMES:
CFTR-mutation screening | 1 year
  CFTR-mutation screening will be carried out in Patients with abnormal results of Sweat Test. Mutation detection analysis will be performed in Next Generation Sequencing method using the genomic DNA extracted from peripheral whole blood.

OTHER OUTCOMES:
Prevelance of CF or CFTR dysfunction | 1 year
  The CF and CFTR dysfunction diagnosis is according to the results of sweat tests combined with CFTR sequencing results. CF is defined as a chloride concentration above 59 mmol/L combined with more than one CFTR mutation, while CFTR dysfunction is defined as a chloride concentration between 30-59mmol/L combined with one or two CFTR mutations.
Microbiology | through study completion, an average of 1 year
  Sputum or bronchoalveolar lavage fluid culture
Bronchiectasis severity Score (BSI) | At baseline and updated once a year for 3 years
  The scale is presented online. It consists of 9 items including Age, BMI(Body Mass Index), % FEV1 Predicted, Previous Hospital Admission in the past 2 years, number of exacerbations in previous year, MRC Breathlessness Score, Pseudomonas Colonisation, Colonisation with other organisms,affected lobes.
  0-4 Mild Bronchiectasis. 5 - 8 Moderate Bronchiectasis. 9 + Severe Bronchiectasis.
Lung function (FEV1 %, FVC %, FEV1/FVC %) | 1 year
  Lung function would be tested by spirometry when patients visit the clinic.
E-FACED score | At baseline and updated once a year for 3 years
  It consists of 6 items including exacerbation history in the past year, % FEV1 predicted, Age, Chronic colonization by Pseudomonas aeruginosa, n° of pulmonary lobes affected,and Dyspnea (measured by mMRC score) mild: 0-3 points, moderate: 4-6 points; and severe: 7-9 points
Comorbidity | At baseline and updated every year for up to 3 years
  Comorbidity would be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-fu Xu, MD, Study Chair — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai pulmonary hospital, Shanghai, Shanghai Municipality, China